FOR IRB USE ONLY
IRB ID #: 201911030
APPROVAL DATE: 06/16/22
RELEASED DATE: 06/17/22
EXPIRATION DATE: N/A

This is a research study conducted by Dr. Jason Newland having to do with adolescent vaccines. The study will test a strategy to increase the use of the Human Papilloma Virus (HPV) vaccine for pre-teens (11 to 13 year-olds). The NIH is funding this study. You may choose to participate or not.

If you agree and complete this survey, you will be volunteering to participate in the research study. As a voluntary participant, you will complete a brief annual survey regarding your beliefs and current practice for HPV vaccination. You will also be asked demographic questions. It will take about 10 minutes to complete each survey. You are free to skip any questions that you prefer not to answer.

There are no known risks from being in this study. You will not benefit personally. However, we hope that others may benefit in the future from what we learn about adolescent vaccination use as a result of this study.

You will not have any costs for being in this research study and you will receive a \$50 Amazon gift card for each completed survey as partial compensation for your time.

We will keep the information you provide confidential by using an ID code number rather than your name on the survey. We will destroy the link between the code number and your name after the study is over. The study team will only use and share your information as talked about in this form.

To further protect your privacy, this research is covered by a Certificate of Confidentiality from the federal government. This means that the researchers can refuse to disclose information that may identify you in any legal or court proceeding or to anyone who is not connected with the research except if:

- there is a law that requires disclosure, such as to report child abuse and neglect, or harm to self or others;
- you give permission to disclose your information, including as described in this consent form; or
- it is used for other scientific research allowed by federal law.

You have the right to share your information or involvement in this study with anyone at any time. You may also give the research team permission to disclose your information to a third party or any other person not connected with the research.

I agree to participate in this survey

- o Yes
- o No